CLINICAL TRIAL: NCT02841904
Title: The Accuracy of Probe-based Confocal Laser Endomicroscopy Versus Conventional Endoscopic Biopsies for the Diagnosis of Superficial Bladder Neoplasia.
Brief Title: The Accuracy of Optic Biopsies Versus Conventional Biopsies for the Diagnosis of Superficial Bladder Neoplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Sami Beji, MD, Medical doctor, Herlev Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-15020548
Record Dates: First submitted 2016-07-07; First posted 2016-07-22 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLE (Other): CLE assessed by the pathologist
  Interventions: Device: Confocal LASER Endomicroscopy
- Biopsy (Active Comparator): Histology assessed by the pathologist
  Interventions: Device: Confocal LASER Endomicroscopy

INTERVENTIONS:
Device: Confocal LASER Endomicroscopy — Patients scheduled for bladder endoscopic surgery under general anesthesia are offered to be included in our study. The suspicious mucosal areas are marked then examined with CLE. Tissue samples are taken based on the usual standard criterias. The samples are evaluated microscopically and compared with the results of the CLE technique. A single surgeon performs all surgeries. Biopsies are anlysed by a pathologist from Herlev and Gentofte Hospital's Pathology Department, which is affiliated CLE- study.
  Other Names: Cellvisio

SUMMARY:
This study evaluates the accuracy of Confocal Laser Endomicroscopy (CLE) in the diagnostic of non-invasive flat and exophytic bladder neoplasia. CLE results are compared to histopathology results.

DETAILED DESCRIPTION:
Confocal Laser Endomicroscopy (CLE) is a technique which during endoscopic examination of the bladder (cystoscopy) gives magnified, microscopic-like images of tissues and cells, by inserting a laser fiber through the cystoscope. CLE aims to target biopsies during cystoscopy and reduce the number of biopsies, and the need for additional cystoscopies i general anesthesia.

This study evaluates the ability of CLE to assess tissue in the bladder. The ability to diagnose normal mucosa, inflammation and tumors of the bladder by the CLE is compared to the histopathological examination of selected tissues (biopsies).

Patients scheduled for cystoscopy with biopsies in general anesthesia are recruited for the study. After standard cystoscopy where suspicious mucosal areas are located and marked, A contrast agent (Fluorescein) is administrated intravenously. CLE fiber is introduced through the cystoscope and the marked mucosal areas are examined by direct contact with the laser fiber. The pathologist assesses the CLE video and registers the results. Biopsies are then taken from the selected, suspicious areas. The results of CLE assessment are compared with the histopathological results.

ELIGIBILITY:
Inclusion Criteria:

* First time Transurethral Resection of Bladder (TURB) for bladder tumors under 3 cm
* Suspicious mucosa / Carcinoma in situ
* Recurrent pTa
* Positive cytology with normal flexible cystoscopy
* Control after Bacille Calmette Guérin (BCG) treatment

Exclusion Criteria:

* Allergy to fluorescein
* Pregnant and lactating women.
* Renal failure (eGFR <20 ml / min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
accordance between CLE and histology in flat bladder tumors | An average of 18 months
  Accordance between confocal laser endoscopy and conventional biopsy according to the evaluation of the pathologist in flat bladder neoplasia
Accordance between CLE and histology in exophytic bladder tumors | An average of 18 months
  Accordance between confocal laser endoscopy and conventional biopsy according to the evaluation of the pathologist in exophytic bladder neoplasia

SECONDARY OUTCOMES:
Accordance between CLE assessed by the surgeon and histology. | An average of 18 months
  Accordance between confocal laser endoscopy and conventional biopsy according to the evaluation of the surgeon in both flat and exophytic bladder neoplasia
Accordance between the per-operative evaluation of CLE of the pathologist and the surgeon | An average of 18 months
  Accordance between the per-operative evaluation of CLE of the pathologist and the surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Sami Beji, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Urology department, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No